CLINICAL TRIAL: NCT00519740
Title: Influence of Nutrition on Nasal and Bronchial Affliction in Patients With Allergy on Grass-Pollen After Low-Dosed Specific Bronchial Provocation
Brief Title: Influence of Nutrition on Nasal and Bronchial Affliction in Patients With Allergy on Grass-Pollen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof Stefan Zielen, Goethe University, Childrens Hospital, Dept of Pulmonology & Allergy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 214/06/FFM
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Bronchial Hyperreactivity; Hypersensitivity; Allergy; Bronchial Asthma
Keywords: grass-pollen; allergy; bronchial hyperreactivity; asthma
MeSH Terms: conditions — Bronchial Hyperreactivity; Hypersensitivity; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: inhalative specific bronchial provocation with grass-pollen

SUMMARY:
The study is meant to observe the influence of nutrition on nasal and bronchial discomfort in patients with allergy on grass pollen after specific bronchial provocation. Therefore, the investigators will record the patients' nutrition habits and measure the blood level of long chained polyunsaturated fatty-acids.

ELIGIBILITY:
Inclusion Criteria:

* age >12 and <45 years
* informed consent
* Known allergy on grass-pollen

Exclusion Criteria:

* age <12 and >45 years
* Clinical asthma requiring regular inhalation
* vital capacity >80%
* FEV1 < 75%
* Chronic disease
* pregnancy
* Inhalative or systemic steroid use
* substance abuse
* incapability of understanding the study's purpose and performance

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
correlation of the blood fatty-acid level and bronchial hyperreactivity, measured as the exhaled NO. | aug 2006 - feb 2007

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, M.D., Ph.D., Principal Investigator — Goethe University, Department of Pulmonology
Locations (1):
- Goethe University, Department of Pulmonology, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Result] Dyerberg J, Bang HO. Lipid metabolism, atherogenesis, and haemostasis in Eskimos: the role of the prostaglandin-3 family. Haemostasis. 1979;8(3-5):227-33. doi: 10.1159/000214314. PMID 511010
- [Derived] Kitz R, Rose MA, Schubert R, Beermann C, Kaufmann A, Bohles HJ, Schulze J, Zielen S. Omega-3 polyunsaturated fatty acids and bronchial inflammation in grass pollen allergy after allergen challenge. Respir Med. 2010 Dec;104(12):1793-8. doi: 10.1016/j.rmed.2010.06.019. Epub 2010 Jul 15. PMID 20637584